CLINICAL TRIAL: NCT06043765
Title: TRUE-GRIT: Reducing Cognitive Impairment in Glioma with Repetitive Transcranial Magnetic Stimulation and Cognitive Strategy Training
Brief Title: Reducing Cognitive Impairment in Glioma with Repetitive Transcranial Magnetic Stimulation and Cognitive Strategy Training
Acronym: TRUE-GRIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linda Douw (Other)
Responsible Party: Sponsor-Investigator, Linda Douw, Associate Professor, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL82233.029.22
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Impairment; Glioma
Keywords: repetitive transcranial magnetic stimulation (rTMS); cognitive strategy training (CST); cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Glioma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive strategy training + real rTMS (Experimental): Verum rTMS to PPC contralateral to the tumor (3000 10Hz pulses at 110% RMT, 30 10-s trains, 30s inter-trial interval, 20 mins total)
  Interventions: Device: real repetitive transcranial magnetic stimulation (rTMS); Behavioral: cognitive strategy training
- Cognitive strategy training + sham rTMS (Sham Comparator): Sham rTMS to PPC contralateral to the tumor (3000 10Hz pulses at 110% RMT, 30 10-s trains, 30s inter-trial interval, 20 mins total).
  Interventions: Device: sham repetitive transcranial magnetic stimulation (rTMS); Behavioral: cognitive strategy training

INTERVENTIONS:
Device: real repetitive transcranial magnetic stimulation (rTMS) — real rTMS -- 3 sessions a week/7 weeks (21 sessions)
  Arms: Cognitive strategy training + real rTMS
Device: sham repetitive transcranial magnetic stimulation (rTMS) — sham rTMS - 3 sessions a week/7 weeks (21 sessions)
  Arms: Cognitive strategy training + sham rTMS
Behavioral: cognitive strategy training — 7 weekly sessions with a trained neuropsychologist.

SUMMARY:
The TRUE-GRIT study will assess the feasibility of a study protocol investigating the efficacy of a combination therapy consisting of cognitive strategy training (CST) and repetitive transcranial magnetic stimulation (rTMS) to reduce cognitive impairment in adult glioma patients. This study is part of the GRIP-project, a project aimed at investigating interventions for improving quality of life in brain tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Histological diagnosis of diffuse glioma (WHO grade 2,3, or 4)
* Subjective cognitive impairment, defined as CFQ-score ≥ 44
* Being able to give informed consent and undergo treatment and measurements based on researchers insight
* Stable disease, i.e. no oncological treatment for ≤ 2 months prior to inclusion; no radiological progression on the most recent MRI, not older than 6 months, and no clinical progression at inclusion
* Stable dosage (for at least 8 weeks) of anti-epileptic medication

Exclusion Criteria:

* Current pregnancy or have given birth less than three months ago
* Current other treatment for cognitive complaints
* Karnofsky performance score <70
* A tumor located in the parietal cortex
* TMS exclusion: implanted medical devices (e.g. pacemaker, deep brain stimulator, cochlear implants, medical infusion device, etc.); metal in the body; sleep deprivation
* MRI exclusion: extreme claustrophobia or metallic objects in or on the body

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients completing intervention and study protocol | Baseline versus directly post-intervention (max. 11 weeks after baseline)
  The feasibility will be assessed by number of patients completing the intervention and obligatory study measurements

SECONDARY OUTCOMES:
Tolerability and side effects of the combination therapy | Weekly during the intervention (7 weeks)
  Tolerability and side-effects will be assessed with an in-house-made questionnaire (with yes/no and open questions)

OTHER OUTCOMES:
Exploratory outcomes: neurocognitive functioning, pre- and post-treatment brain activity, connectivity and network topology. | Baseline versus directly post-intervention (max. 11 weeks after baseline)
  Exploratory parameters are measured as they will be of relevance for a subsequent RCT in case of proven feasibility. Measurements: MRI, MEG, neuropsychological assessment and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Douw, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Centers, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the GRIP project, of which TRUE-GRIT is part of (in Dutch) — https://www.amc.nl/web/research/trials-collaborations/het-grip-programma.htm